CLINICAL TRIAL: NCT04155346
Title: Feasibility and Effectiveness of Prehabilitation in High-risk Surgical Patients
Brief Title: Prehab for Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); MSH-UHN AMO Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Daniel Santa Mina, PhD, Assistant Professor, University of Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-5573
Record Dates: First submitted 2019-10-30; First posted 2019-11-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Surgical Patients; Preoperative Care
Keywords: Exercise; Nutrition; Psychology; Prehabilitation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation hybrid model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facility-based prehabilitation (FBP) (Experimental): Exercise
  * Three supervised exercise training sessions of aerobic and resistance exercises. Includes high-intensity interval aerobic training and whole-body resistance exercises (60 min/session)
  * Specific exercises will also be prescribed to prepare regional and/or compensatory tissues for surgery
  * Exercise session will be supervised by a Registered Kinesiologist/Exercise Physiologist
  Nutrition
  * Participants will receive an individualized nutrition assessment and counselling within the first week of prehabilitation and again in the week prior to surgery
  * All sessions will conducted by a Registered Dietitian (60 min/session)
  * Participants will also receive 20g of protein supplementation daily
  Stress management and behavioural support
  * Participants will be scheduled for a psychoeducation session within the first week of prehabilitation and again in the week prior to surgery
  * All sessions will conducted by a psychologist (60 min/session)
  Interventions: Behavioral: Exercise, nutritional optimization, and psychoeducation
- Home-based prehabilitation (HBP) (Experimental): Exercise
  * Three unsupervised, home-based exercise training sessions of aerobic and resistance exercises. Includes continuous moderate-intensity aerobic training and whole-body resistance exercises (60 min/session)
  * Specific exercises will also be prescribed to prepare regional and/or compensatory tissues for surgery
  * Exercise session will be supervised by a Registered Kinesiologist/Exercise Physiologist
  Nutrition
  * Participants will receive an individualized nutrition assessment and counselling within the first week of prehabilitation and again in the week prior to surgery
  * All sessions will conducted by a Registered Dietitian (60 min/session)
  * Participants will also receive 20g of protein supplementation daily
  Stress management and behavioural support
  * Participants will be scheduled for a psychoeducation session within the first week of prehabilitation and again in the week prior to surgery
  * All sessions will conducted by a psychologist (60 min/session)
  Interventions: Behavioral: Exercise, nutritional optimization, and psychoeducation
- Usual Care (No Intervention): - This group will receive no additional intervention from the routine care.

INTERVENTIONS:
Behavioral: Exercise, nutritional optimization, and psychoeducation — Multimodal prehabilitation including exercise, nutrition, and stress-management delivered via a facility-based or home-based model
  Arms: Facility-based prehabilitation (FBP); Home-based prehabilitation (HBP)

SUMMARY:
Surgical prehabilitation is the process of enhancing one's physical function and mental capacity to enable him/or her to withstand the stressor of surgery. Prehabilitation can be achieved via optimizing physical fitness, nutrition, and psychological health. Studies have shown that prehabilitation may prevent complications during and after surgery, reduce hospital length of stay, and improve postoperative recovery. Despite the growing interest in the field of prehabilitation, little is understood about how to implement prehabilitation an integrated clinical service. This study will examine the effect of a prehabilitation program that includes exercise, psychological, and nutritional optimization that emulates clinical integration pathways. Participants of this study will have a choice of participating in facility-based prehabilitation (FBP) or home-based prehabilitation (HBP) depending on their needs/accessibility to the Toronto General Hospital. Participant outcomes will be measured using standardized fitness testing, self-report questionnaires, and medical record reviews at baseline, one week preoperatively, and at 30 and 90 days postoperatively. A comprehensive assessment of feasibility will also be conducted to better understand facilitators and barriers to clinical integration.

DETAILED DESCRIPTION:
There is growing interest in the role of prehabilitation to reduce surgical risk, attenuate surgery-related deconditioning, and facilitate postoperative recovery. Compared to the postoperative setting, initiating health interventions preoperatively is proposed as an important strategy to improve health outcomes because: i) it targets modifiable risk factors for surgical complications; ii) patients may be more physically and/or psychologically capable of affecting change in health status compared to the early postoperative period; iii) wait times prior to surgery may be several weeks thus representing an opportunity to proactively invest in their recovery; and iv) patients may be sensitized to the importance of adverse health behaviours that may have contributed to the need for surgery (i.e. a 'teachable moment'). The potential benefit of prehabilitation extends beyond potential gains in health from baseline to surgery, but also includes the prevention or attenuation of deconditioning that patients experience during the postoperative period. The findings of recent systematic reviews and meta-analyses assessing the benefits of prehabilitation interventions in surgical patients provide support for their efficacy in improving physical fitness, length of stay, surgical complication rates, and health-related quality of life (HRQOL).

While previous interventional studies have demonstrated promising findings, little is known about how feasible it is to integrate prehabilitation into standard of care for people awaiting surgery. This study intends to employ intervention design features previously shown to be feasible and efficacious and employs a hybrid effectiveness-implementation trial design model to assess feasibility of clinical integration.

ELIGIBILITY:
Inclusion Criteria:

* Planned for surgery at the University Health Network
* Fluent in English
* Referred by their surgeon with indication for prehabilitation as per the surgeon's clinical impression (i.e. higher-than-average risk candidate; marginal candidate for surgery due to limited physiologic reserve; frail; deconditioned; or other reason with explanation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Referral and Enrollment Data | Baseline
  * The number of eligible patients per month who consent for surgery will be ascertained via the preadmission clinic databases.
  * The total number of referrals received from surgeons.
  * The number of patients that agree to participate in the prehabilitation program.
  * Demographics, disease characteristics, and treatment type will be captured for prehabilitation participants
  * Referred patients who decline participation in the study will be compared to all consenting participants using information provided on the referral form
  * For those who fail screening or decline participation, we will log their demographic and reasons for non-participation.
Window of opportunity | Baseline to surgery
  The 'prehabilitation window' will be recorded and is operationally defined as the time from program referral to the date of surgery. We will also describe the total preoperative period (time between consent for surgery and date of surgery) and prehabilitation program duration (time from program initiation to surgery). Each of these periods will be recorded in days.
Intervention adherence and fidelity | Baseline to surgery
  * Adherence for FBP participants will be recorded via attendance to each in-person session. Fidelity and adherence will be further measured by detailed recording of performance on the aerobic and resistance training components of the exercise sessions.
  * HBP participants will be contacted weekly via telephone or email for adherence recording by the research coordinator. A logbook will be used to self-report HBP participants' home-based exercise that contains specific fields to capture all session details.
  * Adherence to stress management and utilization of smoking cessation tools (as required) will be recorded weekly using a logbook within the participant manuals. This includes the number of relaxation sessions per week; compliance with dietary recommendations for dietary behaviours, protein supplementation, and for smokers, the tools used, and the number of times accessed.
Study retention | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  - The frequency of drop-out during program participation will be documented including reasons for drop-out. Descriptive statistics for demographic data and reasons will be used to describe program completers and drop-outs.
Barriers and facilitators | 30-day postoperatively
  Qualitative content analysis on barriers and facilitators for prehabilitation participation and engagement will be conducted using semi-structured interviews. Both participants of prehabilitation and usual care will be asked to participate in interviews via telephone or in-person. To reach saturation for identifying meta-themes within a heterogenous population, sample of has been suggested 15 for the collection of prevalent and more salient ideas.
Safety and adverse events | Baseline to surgery
  Any safety or adverse events related to the prehabilitation intervention will be reported at each in-person session for FBP participants and during weekly telephone calls with HBP participants. Reporting and grading will follow the Common Terminology Criteria for Adverse Events version 5.0.
Economic feasibility (hospital perspective) | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  A cost impact on the perspective of the hospital will be conducted based on primary hospital length of stay, readmission, and readmission length of stay. This will be used to determine cost differences between those that participate in prehabilitation (FBP and HBP) compared to usual care.
Economic feasibility (patient perspective) | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  Patient-perspective costing will be measured by a patient-reported cost-diary. This includes: direct healthcare cost (i.e. visits to the general practice, specialists care, unities applied to prescribed medication); direct non-health care costs (i.e. cost of over-the-counter medication, cost of health activities, hours of paid and unpaid household help, transportation, and value of other out-of-pocket expenses, with specifics on exercise-related expenses)l and indirect costs (i.e. number of days absent from work, days lost from housekeeping, and other daily activities).

SECONDARY OUTCOMES:
Hospital length of stay | Up to 90-days postoperatively
  Postoperative length of stay will be recorded from the patient's medical record. This will be calculated from the date of surgery until to the date of discharge from the hospital and recorded in hours.
Postoperative complications and mortality | Up to 90-days postoperatively
  Complications, including mortality, will follow the Clavien-Dindo classification. Any health event that requires readmission will also be documented.
Changes in aerobic functional capacity | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  Aerobic functional capacity will be measured using the Six-Minute Walk Test (6MWT). Total distance travelled for 6 minutes will be recorded. Measured only in participants of prehabilitation.
Changes in musculoskeletal functional capacity | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  Musculoskeletal functional capacity will be assessed via grip strength. Peak isometric force generated for both arms will be recorded in kg-force. Measured only in participants of prehabilitation.
Changes in body composition | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  Body composition will be measured via bioelectric impedance analysis using mBCA 514 (Seca, Hamburg, Germany). Body fat percentage, fat and fat free mass, impedance, resistance, and phase angle will be recorded. Measured only in participants of prehabilitation.
Changes in HRQOL | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  HRQOL will be measured by Short Form-12 Health Survey (SF-12) and the EuroQol-5 Dimension (EQ5D). Measured only in participants of prehabilitation.
Changes in depression | Baseline, 1 week prior to surgery, 30- and 90-day postoperatively
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9). Measured only in participants of prehabilitation.
Changes in diet | Baseline and 1 week prior to surgery
  Changes in diet and healthy eating practices will be measured by the 3-day diet record. Measured only in participants of prehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Santa Mina, PhD, Principal Investigator — University of Toronto; Ian Randall, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada